CLINICAL TRIAL: NCT04881097
Title: Cognitive Function and Health-related Quality of Life After Neuro-intensive Care: An Observational Multicenter Cohort Study
Brief Title: Cognitive Function and Health-related Quality of Life After Neuro-intensive Care
Acronym: COGNI
Status: Withdrawn | Type: Observational
Why Stopped: Primary Investigator ceased their involvement with study
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kirsten Moller, Professor, Rigshospitalet, Denmark
Other Study IDs: NNF 20OC0064760
Record Dates: First submitted 2021-04-22; First posted 2021-05-11 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Acute Brain Injury; Cognitive Dysfunction; Delirium; Sepsis; Post-traumatic Amnesia; Health-related Quality of Life
Keywords: Acute brain injury after intensive care unit care
MeSH Terms: conditions — Brain Injuries; Cognitive Dysfunction; Delirium; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: no intervention — no intervention

SUMMARY:
The study will provide information on cognitive impairment and Health related quality of life in patients surviving 12 months after acute brain injury, generate a hypothesis of useful variables to predict cognitive impairment or low levels of HRQoL, and potentially inform interventions for the prevention and treatment of cognitive impairment following neuro-ICU stay.

DETAILED DESCRIPTION:
The aim is to 1) measure the frequency and extent of cognitive impairment after acute brain injury at six and 12-months after neuro-Intensive care unit (ICU) admission 2) explore the association between cognitive impairment at six and 12 months after ICU admission with the following potential risk factors: duration of ICU delirium (days), duration of sepsis (days), duration of post traumatic amnesia (days) and the severity of brain injury (initial Glasgow Coma Scale , 3) describe Health related quality of life, functional disability and frailty at six and 12 after ICU admission and 4) explore the association between the functional disability, frailty and health-related quality of life at 12 months after ICU admission

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury
* Spontaneous intracranial hemorrhage
* Ischemic stroke
* An anticipated stay in the neuro-ICU for 48 hours or longer.

Exclusion Criteria:

* Persistent coma defined as Richmond Agitation-Sedation Scale (RASS) -5 to -3 throughout the neuro-ICU stay
* Congenital brain injury
* Suspected pre-existing Cognitive impairment (Informant Questionnaire on cognitive decline in the elderly (IQCODE): 3.3 or more) (regardless of cause)
* Permanent residence outside Denmark
* Inability to communicate in Danish

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with acute brain injury from traumatic brain injury, spontaneous intracranial hemorrhage, or ischemic stroke with a Neuro ICU stay
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Global cognitive function | from baseline to 6 months after ICU admission
  measured by The Repeatable Battery for the Assessment of Neuropsychological Status, Overall score (mean 100; SD=15). Higher scores indicate better cognitive functioning.
Change in Global cognitive function | from baseline to 12 months after ICU admission
  measured by The Repeatable Battery for the Assessment of Neuropsychological Status, Overall score (mean 100; SD=15). Higher scores indicate better cognitive functioning.
Change in Executive function | from baseline to 6 months after ICU admission
  measured by Trail Making Test B, Score indicate time in seconds to complete task, the higher speed (less seconds) indicates higher executive function
Change in Executive function | from baseline to 12 months after ICU admission
  measured by Trail Making Test B, Score indicate time in seconds to complete task, the higher speed (less seconds) indicates higher executive function

SECONDARY OUTCOMES:
Change in Health related quality of life after brain injury | from baseline to 6 months after ICU admission
  measured with a disease specific questionnaire:Quality of Life after Brain Injury overall scale (QOLIBRI-OS). Scores are from 0-100, the higher the score the more quality of life.
Change in Health related quality of life after brain injury | from baseline to 12 months after ICU admission
  measured with a disease specific questionnaire:Quality of Life after Brain Injury overall scale (QOLIBRI-OS). Scores are from 0-100, the higher the score the more quality of life.
Delirium | during the procedure (ICU stay) up to 30 days
  measured by Confusion measured by CAM-ICU or Intensive Care Delirium Screening Checklist (ICDSC).
Change in Disability after head injury/nontraumatic acute brain insults I | from baseline to 6 months after ICU admission
  measured by Glasgow outcome scale extended (GOSE). Scores from 1 to 8, higher scores indicate less disability
Change in Disability after head injury/nontraumatic acute brain insults I | from baseline to 12 months after ICU admission
  measured by Glasgow outcome scale extended (GOSE). Scores from 1 to 8, higher scores indicate less disability
Change in Disability after head injury/nontraumatic acute brain insults II | from baseline to 6 months after ICU admission
  measured by Extended disability rating scale (DRS). Scores from 0 to 29, the higher the score the more disability
Change in Disability after head injury/nontraumatic acute brain insults II | from baseline to 12 months after ICU admission
  measured by Extended disability rating scale (DRS). Scores from 0 to 29, the higher the score the more disability
Change in Frailty | baseline to 6 months after ICU admission
  measured by the Clinical Frailty Scale (CFS). Scale is from 1 to 9 ( the higher score the more frail).
Change in Frailty | baseline to 12 months after ICU admission
  measured by the Clinical Frailty Scale (CFS). Scale is from 1 to 9 ( the higher score the more frail).

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne F Herling, Ph.D, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No